CLINICAL TRIAL: NCT03379805
Title: The Lymphatic Morphology and Function of Fontan-Kreutzer Operated Patients
Brief Title: Lymphatic Function in Patients With a Fontan-Kreutzer Circulation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Fontan17
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Lymphatic Abnormalities; Lymphatic Edema; Univentricular Heart
MeSH Terms: conditions — Lymphatic Abnormalities; Lymphedema; Univentricular Heart

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan-Kreutzer operated patients: Patients with a Fontan-Kreutzer circulation. No interventions are done. (The intervention is the operation done 15-20 years ago)
  Interventions: Diagnostic Test: Near Infrared Fluorescence Imaging; Diagnostic Test: Non-contrast MRI; Diagnostic Test: Strain Gauge Plethysmography
- Healthy Control subjects: Age, gender and weight matched control subjects
  Interventions: Diagnostic Test: Near Infrared Fluorescence Imaging; Diagnostic Test: Non-contrast MRI; Diagnostic Test: Strain Gauge Plethysmography

INTERVENTIONS:
Diagnostic Test: Near Infrared Fluorescence Imaging — The functional state of lymphatics is investigated using near infrared fluorescence imaging, NIRF.
  Other Names: Strain-Gauge Plethysmography
Diagnostic Test: Non-contrast MRI — The anatomy is described using non-contrast MRI.
Diagnostic Test: Strain Gauge Plethysmography — The capillary filtration rate is measured using plethysmography

SUMMARY:
The lymphatics regulate the interstitial fluid by removing excessive fluid. It represents an extremely important step in the prevention of edema. The Fontan-Kreutzer procedure has revolutionized the treatment of univentricular hearts. However, it is associated with severe complications such as protein-losing enteropathy (PLE) and peripheral edema that may involve the lymphatic circulation.

Our hypothesis is that patients with a univentricular circulation have a reduced functionality of the lymphatic vasculature, which predisposes them to developing complications such as edema and PLE.

The functional state of lymphatics is investigated using near infrared fluorescence imaging, NIRF. The anatomy is described using non-contrast MRI and the capillary filtration rate is measured using plethysmography.

DETAILED DESCRIPTION:
Background:

The lymphatics regulate the interstitial fluid by removing excessive fluid. It represents an extremely important step in the prevention of edema. The Fontan-Kreutzer procedure has revolutionized the treatment of univentricular hearts. However, it is associated with severe complications such as protein-losing enteropathy (PLE) and peripheral edema that may involve the lymphatic circulation.

Hypothesis:

Patients with a univentricular circulation have a reduced functionality of the lymphatic vasculature, which predisposes them to developing complications such as edema and PLE.

Material and Methods:

The functional state of lymphatics is investigated using near infrared fluorescence imaging, NIRF. The anatomy is described using non-contrast MRI and the capillary filtration rate is measured using plethysmography. The study population is patients with Fontan-Kreutzer circulation operated at Aarhus University hospital. Exclusion criteria is BMI>30 and age (years) < 18. The Fontan-Kreutzer group will be compared with an age, gender and weight matched control group of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Fontan-Kreutzer circulation

Exclusion Criteria:

* BMI>30,
* Age<18
* Mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients born with an univentricular heart, who surgically is corrected with a Fontan-Kreutzer Circulation
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-04-25 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Pumping pressure | 1 hour
  Occlusion of lymphatic flow by inflating a cuff (Hokanson E20 Rapid cuff inflator, Hokanson AG101 air source) to 70mmHg and then reducing the pressure with 5mmHg each 5th minute. The highest pressure under which the fluorescent dye is able to cross the inflatable cuff is labelled Ppump.
Contraction Frequency | 6 min
  Contraction frequency in vessels in the main drainage pathway of the legs (ventromedial bundle) as well as vessels draining the area behind the medial malleolus.
Refill time | 20 min
  The time it takes for a 10 cm long vessel to refill after emptying the vessel with massage
Velocity | 6 min
  The velocity measured in cm/s for a packet of lymph moving from one region of interest (ROI) to another through atlas a 5 cm straight vessel
Capillary Filtration Rate | 25 min
  A 5-step 20-min venous congestion protocol will be used to measure capillary filtration. The capillary filtration rate (µl·100 ml-1 ·min-1 ) is measured as the slope of the time-volume change (%) curve at steady state at the end of each pressure phase.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, MD, PhD, Dr.Med, Principal Investigator — Aarhus University Hospital, Department of Cardiothoracic and Vascular Surgery

REFERENCES:
- [Derived] Mohanakumar S, Telinius N, Kelly B, Lauridsen H, Boedtkjer D, Pedersen M, de Leval M, Hjortdal V. Morphology and Function of the Lymphatic Vasculature in Patients With a Fontan Circulation. Circ Cardiovasc Imaging. 2019 Apr;12(4):e008074. doi: 10.1161/CIRCIMAGING.118.008074. PMID 30943769